CLINICAL TRIAL: NCT04992377
Title: A Multicenter Phase 2 Study of R-EPOCH in Combination With Ibrutinib for Patients With Classical Richter Transformation of Chronic Lymphocytic Leukemia
Brief Title: R-EPOCH in Combination With Ibrutinib for Patients With Classical RT of CLL
Acronym: BDHRT001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Principal Investigator, Tingyu Wang, associate chief physician, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHBDH-IIT2021015
Record Dates: First submitted 2021-07-16; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Richter Transformation
Keywords: Richter transformation; chronic lymphocytic leukemia; R-EPOCH; Ibrutinib; Therapeutics
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- R-EPOCH plus IBR for RT (Experimental)
  Interventions: Drug: R-EPOCH in Combination With Ibrutinib

INTERVENTIONS:
Drug: R-EPOCH in Combination With Ibrutinib — Induction:
  (21-day per cycle) Ibrutinib:420mg given orally , once daily.
  Details of R-DA-EPOCH are as follows:
  Rituximab: 375 mg/m2 given intravenously (IV) on day 0 Etoposide: 50 mg/m2 given CIV from day 1-4 Doxorubicin: 10 mg/m2 given CIV from day 1-4 Vincristine: 0.4 mg/m2 given CIV from day 1-4 Cyclophosphamide: 750 mg/m2/day IV on day 5 Prednisone: 60 mg/m2 given orally bid on days 1-5. Patients who achieve CR after 4 cycles enter the consolidation treatment ; Patients with PR after 4 cycles would receive another 2 cycles of R-EPOCH + ibrutinib induction therapy, they could enter the consolidation treatment if they achieve CR ,withdrawn from the study if they achieve ≤ PR; Patients with SD/PD after 4 cycles of treatment are withdrawn from the study.
  Consolidation:
  2 cycles of R-EPOCH + Ibrutinib (dose as before) treatment
  Maintenance:
  Ibrutinib 420 mg/day for 24 months or until disease progression or intolerable toxicity

SUMMARY:
This is an investigator-initiated Phase 2 study, which combines R-EDOCH with Ibrutinib to treat patients with Ritcher Transformation in consideration of DLBCL and CLL components both could being targeted at the same time. The investigator will observe the 2-year overall survival rate of this regimen for RT and explore the new regimen for RT in the novel drugs era, which aims to improve the efficacy and prolong survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. ECOG 0-2
3. Confirmed Richter transformation, whether or not previously treated
4. Unexposed to BTKi, or discontinue BTKi more than 1 year (due not to toxicity or ineffectiveness)
5. No serious liver, kidney, heart and other complications; including: a. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal (ULN); b. total bilirubin (TBIL) ≤ 1.5 times the ULN; c. serum creatinine (Cr) ≤ 2 times the ULN, or glomerular filtration rate ≥ 40ml/min; d. LVEF > 50% determined by echocardiography; e. no arrhythmia and active heart disease, such as coronary heart disease, myocardial infarction, etc
6. The patient agreed to participate and signed the informed consent form

Exclusion Criteria:

1. Major surgery within 4 weeks prior to first dose of ibrutinib
2. Require receiving anticoagulation with warfarin or equivalent Vitamin K antagonists; Requires treatment with a strong CYP3A4/5 inhibitor
3. Require corticosteroid , anti-cancer drugs, immunomodulatory or Chinese medicine for other medical conditions
4. Pregnant or lactating women
5. History of prior malignancy
6. Currently active clinically significant cardiovascular disease
7. Uncontrolled active systemic fungal, bacterial, viral, or other infection
8. Known history of human immunodeficiency virus (HIV) or active infection with Hepatitis B or Hepatitis C
9. History of stroke or intracranial hemorrhage prior to randomization
10. Other conditions that is unfit for the clinical trial in the investigator' opinion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival rate (OS) | 2 years
  Defined as the time interval from enrollment to death of patients in the intent-to-treat population (ITT). If the patient is alive or death of the patient is unknown, the date of death will be the latest time point at which the patient was known to be alive.

SECONDARY OUTCOMES:
Complete response rate (CRR) | 1 month after completion of consolidation therapy
  Defined as the percentage of subjects who achieved CR after treatment in the per-protocol population as well as in the intent-to-treat population.
Overall response rate (ORR) | 1 month after completion of consolidation therapy
  Defined as the percentage of subjects who achieved CR + PR after treatment in the per-protocol population and the intention-to-treat population.
Progression-free survival (PFS) | 2 years
  Defined as the time interval from enrollment to disease progression or death, whichever occurred first, for patients in the intent-to-treat (ITT) population. If there is no progression or time of disease progression is not recorded at the time of withdrawal from the trial, the date of the last examination will be used as the endpoint date.
Minimal residual disease (MRD) negative rate | 1 month after completion of consolidation therapy
  For patients with bone marrow invasion, on the basis of CR, multicolor flow cytometry detects that tumor cells account for the proportion of nuclear cells, and < 0.01% are MRD negative.
Toxic side effects | 3 years
  Non-hematologic toxicity was evaluated according to NCI CTCAE 5.0 criteria; hematologic toxicity was evaluated according to NCI CLL 2018 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Tingyu Wang, Principal Investigator — State Key Laboratory of Experimental Hematology, National Clinical Research Center for Hematological Disorders, Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (11):
- China (11):
  - Peking university Third Hospital, Beijing, Beijing Municipality
  - The second hospital of Hebei medical university, Shijiazhuang, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The second Xiangya hospital of central south university, Changsha, Hunan
  - The First affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First affiliated hospital of China medical university, Shenyang, Liaoning
  - Shandong Cancer Hospital and Institute, Shandong First Medical University and Shandong Academy of Medical Sciences, Jinan, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Tianjin university general hospital, Tianjin, Tianjin Municipality